CLINICAL TRIAL: NCT06582043
Title: Evaluation of the Efficacy and Tolerance of Two Cosmetic Products in Subjects Presenting With Rosacea Treated With Topical Treatment
Brief Title: Evaluation of the Efficacy and Tolerance of Two Cosmetic Products in Subjects With Rosacea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NAOS Argentina S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RC2024/SCARCr/AR-BR
Record Dates: First submitted 2024-08-15; First posted 2024-09-03 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2024-08

CONDITIONS: Rosacea; Redness; Telangiectasia; Flushing; Pustular Acne; Papule Pruritic
Keywords: Rosacea
MeSH Terms: conditions — Rosacea; Erythema; Telangiectasis; Flushing

STUDY DESIGN:
Intervention Model Description: Multicentric and double-blind randomised comparative clinical study in Argentina and Brazil. Under dermatological and ophthalmological control
Who Masked: Participant, Care Provider, Investigator
Masking Description: Randomization for product allocation will consider: number of papules/pustules (<3, ≥3), age (18-35, 35-50, >51), phototype (I-III and IV), sun protector (always, sometimes, never)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SCARCr tester 1 (Active Comparator): The subjects will apply the product concomitantly with the topical medical treatment for 56 days, followed by 28 days applying the SCARCr tester 1 alone.
  Instructions for topical medical treatment and study product application:
  1. Application of the topical treatment (metronidazole twice daily, morning and night, or ivermectin daily at night)
  2. After 5 minutes, application of the study product starting on the eye area followed by the whole face and neck, twice a day, morning and evening.
  Subjects must keep their usual habits during the clinical study (hygiene products, sunscreen, make-up). If the application of sunscreen
  Interventions: Other: SCARCr tester 1; Other: Placebo
- SCARCr tester 2 (Placebo Comparator): The subjects will apply the product concomitantly with the topical medical treatment for 56 days, followed by 28 days applying the SCARCr tester 2 alone.
  Instructions for topical medical treatment and study product application:
  1. Application of the topical treatment (metronidazole twice daily, morning and night, or ivermectin daily at night)
  2. After 5 minutes, application of the study product starting on the eye area followed by the whole face and neck, twice a day, morning and evening.
  Subjects must keep their usual habits during the clinical study (hygiene products, sunscreen, make-up). If the application of sunscreen
  Interventions: Other: SCARCr tester 1; Other: Placebo

INTERVENTIONS:
Other: SCARCr tester 1 — Twice daily
Other: Placebo — Twice daily

SUMMARY:
Multicentric and double-blind randomised comparative clinical study in Argentina and Brazil. Under dermatological and ophthalmological control 4 visits: inclusion [Day(D)0], D28, D56, D84 Ethical committee required.

DETAILED DESCRIPTION:
Primary objective:

To evaluate the efficacy of two cosmetic products (SCARCr tester 1 and SCARCr tester 2) in association to the topical medical treatment (Ivermectin or Metronidazole) in supporting the improvement of persistent redness due to rosacea and in soothing discomfort sensations, under dermatological and ophthalmological control.

Secondary objectives:

To evaluate the cutaneous and ocular tolerance of two cosmetic products in subjects presenting with rosacea under treatment with topical Ivermectin or Metronidazole for 56 days, and 28 days after applying the cosmetic products alone. To evaluate the efficacyof two cosmetic products through clinical evaluation of the symptoms related to rosacea after 56 days of concomitant use of the cosmetic product with the topical medical treatment, and 28 days after applying the cosmetic products alone. To evaluate the efficacyof two cosmetic products through instrumental measurements of redness after 56 days of concomitant use of the cosmetic product with the topical medical treatment, and 28 days after applying the cosmetic products alone. To evaluate the evolution of the quality of life of the subjects over the period of use of the association of the topical medical treatment with the cosmetic products (56 days) and 28 days after applying the cosmetic products alone. To evaluate the immediate and long-lasting eCicacy and cosmetic qualities of the cosmetic products based on self-assessment questionnaires by the subjects. To compare the two products tolerance and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Subject with facial vascular rosacea with flushing, permanent redness, telangiectasias and at least 3 papules and/or pustules (this last criterion for at least 10 subjects per group)
* Subject starting local treatment for rosacea (Ivermectin or metronidazole)
* Female aged 18 to 65 years old,
* Subject of all types of skin
* Subject of I to IV phototype.
* Subject accepting not to use any type of facial skin care other than the study product
* Subject willing to keep their usual habits and products (hygiene products, sunscreen, and make-up, if applicable)
* Subject willing to avoid sun exposure during the study period
* Subject willing to actively participate in the study and to come to the scheduled visits
* Subject that has signed informed consent

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Subject showing cutaneous marks on the experimental areas, which could interfere with the assessment of skin reactions (pigmentation troubles, scar elements, over-developed pilosity, ephelides and naevi in too great quantity, sunburn)
* Subject with documented allergy or reactivity to products of the same category than the tested one
* Subject with documented allergies to study product components
* Subject with history of malignant melanomas (Dubreuilh melanosis…)
* Subject with unbalanced hormonal treatment
* Subject with forecast of initiation of a hormonal treatment or change of the usual hormonal treatment during the study period
* Subject with forecast of sun or UVA exposure (UV lamps) during the study period
* Subject not willing to use sun protective clothes orhat if exposed to the sun
* Subject not willing to respect the methods of use of the treatment, study product and sunscreen
* Subject with anti-ageing or aesthetic treatment during the last 6 months: botox or botox like products, peelings, plastic surgery, hyaluronic acid treatment, Plasma Rich Platelets treatment, or any other specific treatments prone to change the skin aspect
* Subject with antibiotic, anti-allergic, anti-inflammatory treatment or treatment with patent medicines containing Vitamin A acid or its derivatives within 4 weeks and during the study (if therapeutic requirement: exclusion foreseen),
* Subject with systemic disorder: cardiovascular, pulmonary, digestive, neurologic, psychiatric, genital, urinary, haematological, endocrine
* Subject presenting chronic diseases with impact on skin
* Subject who has undergone a bilateral mastectomy with lymph node removal, a unilateral mastectomy with lymph node removal within the last year, or a bilateral axillary lymph node removal,
* Subject with a history of immune deficiency or auto-immune disease, treated for malignancy within 6 months prior to enrolment or who are currently under treatment for asthma or diabetes, forecast of vaccination during the test period or last vaccination within 3 weeks before the study.
* Subject receiving local treatment for rosacea (cyclins, isotretinoin) or who has undergone local active treatment for rosacea (erythromycin, metronidazole, benzoyl peroxide, ivermectin) within 4 weeks before inclusion in the study
* Subject who has had oral treatment with metronidazole or cyclins within 4 weeks before inclusion in the study
* Subject who has had topical or oral anti-inflammatory and/or antiallergy treatment (corticosteroid, antihistamine, anti-inflammatory drugs, immunosuppressives) within 4 weeks before inclusion in the study
* Subject who has had oral treatment with retinoids within 2 months before inclusion in the study
* Subject currently receiving electrocoagulation or laser treatment for telangiectasia

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2024-05-16 (Actual); Primary Completion 2025-01-09 (Actual); Study Completion 2025-02-06 (Actual)

PRIMARY OUTCOMES:
Investigator Global Assessment (IGA) | Day 0- Day 28- Day 56- Day 84
  To evaluate the efficacy of two cosmetic products (SCARCr tester 1 and SCARCr tester 2) in association to the topical medical treatment (ivermectin or metronidazole) in supporting the improvement of persistent redness due to rosacea and in soothing discomfort sensations, under dermatological and ophthalmological control (scoring scale from better to worse value: clear, minimal, mild and mild to moderate).

SECONDARY OUTCOMES:
Cutaneous and ocular tolerance | Day 0- Day 28- Day 56- Day 84
  Collection of adverse events

OTHER OUTCOMES:
Evolution of the quality of life RosaQoL (Rosacea Quality of Life) questionnaire | Day 0- Day 28- Day 56- Day 84
  Scoring scale from better to worse value: never, rarely, sometimes, often and always. Minimum value: never; Maximun value: always.
Evolution of the quality of life Mood Pict | Day 0- Day 28- Day 56- Day 84
  Scoring scale from better to worse value: not at all, lightly, moderate, a lot and extremely.
Evolution of the quality of life Feel Pict questionnaires | Day 0- Day 28- Day 56- Day 84
  Scoring scale from better to worse value; low and high.
Evaluate the immediate and long-lasting eficacy and cosmetic qualities | Day 0- Day 28- Day 56- Day 84
  Self-assessment questionnaires by the subjects (scoring scale from better to worse value: totally agree, agree, disagree and totally disagree).

CONTACTS AND LOCATIONS:
Locations (2):
- Cirec Latam, Ciudad Autónoma de Buenos Aire, Argentina
- MEDCIN, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No